CLINICAL TRIAL: NCT01386918
Title: A Randomized Double-Blind Sham-Controlled Trial of Transcranial Magnetic Stimulation for Refractory Auditory Hallucinations in Schizophrenia
Brief Title: Repetitive Transcranial Magnetic Stimulation for Refractory Auditory Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Dr., Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 127/2003
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Refractory Schizophrenia
Keywords: Hallucinations; Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Hallucinations; Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low frequency left (LFL) sided rTMS (Experimental): LFL rTMS was administered at an intensity of 115% resting motor threshold at 1HZ for 20 minutes. The treatment targeted the left temporoparietal cortex (TPC).
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Priming stimulation (Experimental): Priming stimulation was administered as follows: 10 minutes of 6 Hz at 90% resting motor threshold (RMT) administered to the left temporoparietal cortex followed by 10 minutes of 1 Hz stimulation at 115% RMT.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham Control (Sham Comparator): Sham stimulation was applied with identical parameters to those for the LFL condition but with the coil angled at 90 degrees off the scalp in a single wing tilt position.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — The treatment involves the administration of a magnetic field applied to a specific area of the brain.
  Other Names: Magstim Rapid (Magstim Company Ltd., Wales, UK)

SUMMARY:
Studies using repetitive transcranial magnetic stimulation (rTMS) as a treatment for refractory auditory hallucinations (AH) in schizophrenia have shown promise. The majority of studies have examined the effect of low frequency left-sided stimulation (LFL) (i.e., 1 Hz) to the temporal parietal cortex (TPC). Priming stimulation (6 Hz) prior to LFL stimulation (hereby simply referred to as priming) has been shown to enhance the neurophysiological effects of LFL rTMS alone and, as such, may lead to greater attenuation of AH. Therefore, this study evaluated the efficacy of priming rTMS and LFL rTMS, compared to sham, applied to the TPC in patients with schizophrenia experiencing refractory auditory hallucinations (AH).

ELIGIBILITY:
Inclusion Criteria:

* voluntary and capable to consent based on the subject's ability to provide a spontaneous narrative description of the key elements of the study
* have a diagnosis of Schizophrenia or Schizoaffective Disorder as confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV)
* between the ages of 18 and 65
* meet criteria for AH of at least moderate severity based on the Positive and Negative Symptom Scale (PANSS)
* willing to keep the dose of antipsychotic stable for the duration of the study
* meet criteria for medication resistance, defined as daily AH despite 2 adequate 6-week trials of at least 2 antipsychotic medications and including 1 atypical antipsychotic medication. An adequate trial is defined as a daily dose of 1000 chlorpromazine equivalents for typical antipsychotics medications and the following dosages for atypical antipsychotic medications: risperidone 6 mg, olanzapine 15 mg, quetiapine 500 mg, clozapine 300 mg.

Exclusion Criteria:

* DSM-IV history of alcohol and/or substance abuse in past month, or alcohol and/or substance dependence in the last 6 months
* presence of concomitant major, unstable medical or neurologic illness, or a history of seizures
* are pregnant
* have received rTMS for any reason in the past
* have had a dose change of usual psychotropic medications in the 4 weeks preceding study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2004-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Psychotic Symptoms Rating Scale (PSYRATS) | 4 weeks
  The primary outcome for this study was response (dichotomous outcome), defined as a 30 percent reduction in the composite score derived from the frequency, duration, loudness and content items of the hallucinations subscale of the Psychotic Symptoms Rating Scale (PSYRATS)

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale - Global | 4 weeks
  response on the global PANSS (30% reduction), PANSS global scale change
Positive and Negative Symptom Scale - Positive subscale | 4 weeks
  response on the positive scale of the PANSS (30% reduction), PANSS positive scale change
Hallucination Change Scale | 4 weeks
  response on the HCS (score < 5)
Auditory Hallucination Rating Scale (AHRS) | 4 weeks
  response on the AHRS and change over time in the AHRS.

CONTACTS AND LOCATIONS:
Overall Officials: Z J Daskalakis, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Blumberger DM, Christensen BK, Zipursky RB, Moller B, Chen R, Fitzgerald PB, Daskalakis ZJ. MRI-targeted repetitive transcranial magnetic stimulation of Heschl's gyrus for refractory auditory hallucinations. Brain Stimul. 2012 Oct;5(4):577-85. doi: 10.1016/j.brs.2011.12.002. Epub 2012 Feb 22. PMID 22410480
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research